CLINICAL TRIAL: NCT06586398
Title: A Pilot Randomized Trial of rTMS for Fatigue and Brain Fog and Neuropsychiatric Symptoms of Long-COVID.
Brief Title: A Pilot rTMS Trial for Neuropsychiatric Symptoms of Long-COVID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-000555
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Long Covid-19; PASC Post Acute Sequelae of COVID 19; Brain Fog; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; Fatigue | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and investigators and outcomes assessors will be blind to the assignment to active or sham rTMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active rTMS (Active Comparator): The rTMS magnet will be set to active stimulation without the knowledge of treating doctors or research team. Only one technician will know the randomization list assignment and will adjust the settings. rTMS treatment will include rTMS to the left dorsolateral prefrontal cortex (DLPFC), followed by rTMS to left primary motor cortex (M1).
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): The rTMS magnet will be set to sham stimulation without the knowledge of the treating doctors or the research team.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Participants will be randomized to 15 sessions of double-blind multi-target rTMS treatment (active vs sham) and then will receive only open-label active stimulation for another 15 sessions. Each session will include rTMS to the left dorsolateral prefrontal cortex (DLPFC), followed by rTMS to left primary motor cortex (M1).
  Other Names: repetitive transcranial magnetic stimulation

SUMMARY:
This is a pilot randomized trial of rTMS for symptoms of fatigue and brain fog, and other neuropsychiatric symptoms of Long-COVID (Post-COVID, post-acute sequelae of COVID-19 infection, PASC). Twenty participants diagnosed with Long-COVID and recruited from the UCLA Long-COVID clinic will be randomized to receive active rTMS versus sham stimulation for 15 treatments followed by another 15 open-label rTMS treatments. Investigators will compare the safety and tolerability of rTMS vs Sham and examine within-group changes in symptoms of fatigue, sleep, pain, mood, and subjective and objective cognitive impairment. This project will provide information and pilot data for future larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Prior hx of PCR confirmed COVID-19 infection. Determined by the PI or participant's physician.
3. Subsequent development of post-acute neuropsychiatric symptoms with fatigue and brain fog as primary outcomes
4. USE of Psychotropic medications
5. Stable on psychotropic medications for 4+ months
6. Confirmed diagnosis of Long COVID
7. Subjects are willing and able to adhere to the treatment schedule and required study visits

Exclusion Criteria:

1. Mentally or legally incapacitated or unable to give informed consent
2. MOCA < or = 24
3. Infection of poor skin condition over the scalp where the rTMS device will be positioned
4. Pregnancy: Female participants will be tested for pregnancy at baseline and agree to use a medically acceptable form of birth control throughout the study, for women younger than 60.
5. Lifetime history of diagnosed bipolar disorder; psychosis, such as schizophrenia, schizophreniform, or schizoaffective disorder; intellectual disability (intellectual developmental disorder); organic brain damage; or suicide attempts in the past 24 months.
6. Severe MDD with suicidality of Psychosis- excluded
7. As-needed use of benzodiazepines and beta-blockers will be permitted but discouraged during assessment days.
8. Current abuse or dependence on alcohol or any illicit drug of abuse (disorder in last 6 months). Any recent use of cocaine or opiates will also be exclusionary.
9. Participants with asthma or with a history of serious, uncontrolled medical illness or instability (including significant cardio-pulmonary disease, organic brain including significant cardio-pulmonary syndrome, pre-existing dementia, seizure disorder, cerebrovascular disease, and diabetes)
10. Taking medications known to lower seizure thresholds (Clozaril/ Wellbutrin)
11. Neurological conditions that include epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, having a history of repetitive or severe head trauma, or primary or secondary tumors in the central nervous system.
12. Presence of an implanted metallic and magnetic-sensitive medical device present in the body scan, including but not limited to a cochlear implant, infusion pump, implanted cardioverter defibrillator, pacemaker, vagus nerve stimulator, aneurysm clip, metal prosthesis, or metal aneurysm clips or coils, staples, or stents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Tolerability as measured by Safteesi survey | Baseline, after every 5th treatment, through study completion, an average of 12 weeks.
  Safteesi is an instrument that assesses any new symptom(s) that participants developed since starting the clinical study.
Safety profile and adverse events | Baseline, after every 5th treatment, through study completion, an average of 12 weeks.
  Study patients will be monitored weekly for the occurrence of adverse events.

SECONDARY OUTCOMES:
Subjective Cognitive impairment assessed by Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | Baseline, after every 5th treatment, through study completion, an average of 12 weeks.
  MISC is a brief 10-item survey that measures perceived cognitive function. The MISCI is normally distributed and has low rates of ceiling and floor effects, excellent internal consistency, and good construct validity in correlation with other measures.
Fatigue assessed by Fatigue Severity Scale (FSS) | Baseline, after every 5th treatment, through study completion, an average of 12 weeks.
  The FSS is a nine-item, self-report instrument designed to assess fatigue as a symptom of different chronic conditions and disorders. The scale addresses fatigue's effect on daily functioning and its relationship to motivation, physical activity, work, family, and social life. Participants will rate the ease with which they are fatigued and the degree to which the symptoms pose a problem.
  Scoring uses a scale that ranges from 1 (completely disagree) to 7 (completely agree) to indicate agreement with the nine statements about fatigue.
Physical and mental health assessed by PROMIS-29 | Baseline, through study completion, an average of 12 weeks.
  The PROMIS-29 measures pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items for each domain.
Alzheimer's Disease Assessment Scale (ADAS-Cog) | Baseline through study completion, an average of 12 weeks.
  Cognitive performance will be assessed by ADAS-Cog
Fatigue assessed by VAS for Fatigue Questionnaire | Baseline, after every 5th treatment, through study completion, an average of 12 weeks.
  VAS is a one-question self-report survey that asks "How much fatigue are you having now?" on a scale of 0 (no fatigue) to 10 (worst possible fatigue).
DKEFS CW | Baseline through study completion, an average of 12 weeks.
  Verbally mediated processing speed and executive functioning will be assessed using the DKEFS Color Word Test.
Verbal Fluency test | Baseline through study completion, an average of 12 weeks.
  The Verbal Fluency test will be used to assess global cognitive abilities.
DKEFS Trailmaking A,B | Baseline through study completion, an average of 12 weeks.
  Speed for attention, sequencing, mental flexibility, visual search, and motor functioning will be assessed by the DKEFS Trailmaking tests.
Test of Premorbid Functioning (TOPF) | Baseline
  TOPF will be used to estimate pre-morbid cognitive and memory functioning.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline through study completion, an average of 12 weeks.
  RBANS story memory subtest is used to assess immediate memory.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline through study completion, an average of 12 weeks.
  RBANS story recall subtest will be used to assess delayed memory
Repeatable Battery for the Assessment of Neuropsychological (RBANS) | Baseline through study completion, an average of 12 weeks.
  Processing speed, short-term visual memory, psychomotor speed, cognitive flexibility, concentration, and motivation will be assessed by RBANS Coding subtest.
DKEFS CWI | Baseline through study completion, an average of 12 weeks.
  Selective attention, cognitive flexibility, and processing speed will be assessed by the DKEFS Color Word Interference test.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States